CLINICAL TRIAL: NCT02816229
Title: Endobronchial Valves in Inoperable Patients With Life-threatening Haemoptysis Refractory to Bronchial Artery Embolisation
Brief Title: Endobronchial Valves in Inoperable Patients With Haemoptysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Dr Brian Allwood, Dr, University of Stellenbosch
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N10/11/386
Record Dates: First submitted 2016-06-23; First posted 2016-06-28 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Haemoptysis
Keywords: Haemoptysis; Aspergillus; Endobronchial valve; Interventional pulmonology; Tuberculosis
MeSH Terms: conditions — Hemoptysis; Tuberculosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insertion of endobronchial valve (Experimental): Patients in this group will have one or more EBV inserted into the relevant lung regions to manage the haemoptysis via flexible bronchoscopy.
  Interventions: Device: Insertion of endobronchial valve
- Best care (No Intervention): Patients will receive best medical care.

INTERVENTIONS:
Device: Insertion of endobronchial valve — One or more endobronchial one- way valves will be inserted into the appropriate lung regions
  Arms: Insertion of endobronchial valve

SUMMARY:
Massive haemoptysis is a life-threatening condition which is commonly seen in patients who have previously had pulmonary tuberculosis. Various treatment options exist such as bronchial artery embolisation (BAE) or surgical resection of the affect lung region. However, BAE is not considered curative as there is often recurrence of haemoptysis. Furthermore, not all patients will be deemed suitable for surgical resection, leaving them with very few treatment options. A possible alternative intervention is the insertion of an endobronchial valve (EBV). It is speculated that blood will collect distal to the one way valve and a thrombus will be formed. There is currently no data describing the use of EBV for the treatment of massive haemoptysis. This RCT aims to explore the use and efficacy of EBV in the management of massive haemoptysis.

DETAILED DESCRIPTION:
Massive haemoptysis commonly occurs in patients who have had tuberculosis. While surgical resection of the affected lung segment can be curative, a large majority of patients may not qualify for surgical intervention for a number of reasons. This leaves them with few options to manage their haemoptysis.

Many patients at Tygerberg Hospital have severely reduced cardiopulmonary reserves secondary to multiple episodes of pulmonary Tuberculosis and often present either a unilateral largely destroyed lung or bilateral disease, which make them unsuitable for surgery. For these unfortunate patients who do not qualify for surgery or repeat BAE, practically no treatment options exist, and a significant proportion die in hospital or after discharge from a recurrent episode of massive haemoptysis. For these patients the only option may be to block the bleeding bronchus (identified by the previous BAE or during bronchoscopy) with a balloon catheter (Fogarty catheter) or placement of haemostatic gauze or gel. All these procedures are, however, of limited benefit. Using a blocking device which could be deployed and left in place permanently or be removed if needed has become a new therapeutic concept. Dutau and colleagues reported the successful use of the endoscopic placement of a silicone Spigot in a 39-year-old-woman with massive haemoptysis which prevented alveolar inundation preceding and during the time of bronchial artery embolisation.

Our institution has a long standing experience in massive haemoptysis, clinically and scientifically. We evaluate about 80-100 patients with life threatening haemoptysis a year. Furthermore, we were involved in an early emphysema trial using the IBVEBV® (Intra-Bronchial Valve) of Spiration and have, therefore, the necessary experience with the valve implantation technique.

No data are available regarding the potential clinical use of endobronchial valves in patients with recurrence of haemoptysis after BAE in patients who are not candidate for surgery or BAE.

This study aims to investigate the use, therapeutic benefit and safety of IBV Zephyr® valves in inoperable patients with haemoptysis not responding to BAE or in cases where BAE is not considered feasible.

This is a prospective randomised intervention-control study, with patients allocated to either best medical care (control) or endobronchial valve (intervention) groups. The valves will be inserted via flexible bronchoscopy into the affected lung regions. The primary outcome measure is the time to resolution of massive haemoptysis. Secondary outcomes will include physical and lung function and the occurrence of complications resulting from the insertion of the EBV.

Statistical analysis will be performed blinded to patient grouping by a statistician, and both univariate and multivariate analyses will be performed using the appropriate parametric and non-parametric tests. Appropriate tests for categorical data (e.g. Chi-squared test) and continuous data (e.g. Kruskal-Wallis, and ANOVA) will be used. Logistic and linear regression modelling will be used for certain outcomes, and multivariate analysis will be performed using stepwise regression modelling and full modelling where appropriate.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Written informed consent
* Current or previously documented admission to hospital with large volume haemoptysis (>200ml/24hour); or haemoptysis with haemodynamic compromise (SBP < 100mmHg for 15 minutes) or requiring fluid resuscitation; haemoptysis requiring intubation or deemed life-threatening by attending clinicians.
* The cause of haemoptysis must be due to severe underlying lung destruction/ bronchiectasis, post-tuberculous lung damage or the presence of an aspergillomata.
* Primary bronchial artery embolisation not considered technically possible* or failed (defined as ongoing haemoptysis of at least 100 ml per day for 7 days or more, cumulative blood loss of > 200 ml / 24 hours, or any volume resulting in a systolic blood pressure < 100 mmHg for 15 minutes or necessitating resuscitation with vasopressors during a period of 30 days after BAE) and repeat BAE not considered feasible*
* Lung resection not possible because of poor cardiopulmonary reserves (as defined by the current ERS/ESTS clinical guidelines28, independently reviewed by a team of consisting of a thoracic surgeon, pulmonologist and anaesthesiologist who will need to in absolute agreement on inoperability and/or lack of cardiopulmonary reserve)

Exclusion Criteria:

* Haemodynamic instability (defined as SBP< 90mmHg requiring ongoing fluid resuscitation or inotropic support)
* Patients necessitating mechanical ventilation because of respiratory failure or airway management
* Active tuberculosis
* High clinical suspicion of lung carcinoma
* Any other condition, which in the opinion of the investigators, places the subject at increased risk for bronchoscopy and EBV placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Rate of termination of haemoptysis | 1 year

SECONDARY OUTCOMES:
Time to recurrence of haemoptysis | 1 year
Improvement in exercise performance | 1 year
Improvement in lung function | 1 year
Recurrence of infection/tuberculsis | 1 year
EBV related complications | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Brian Allwood, MBChB, PhD, Study Chair — University of Stellenbosch

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van den Heuvel MM, Els Z, Koegelenberg CF, Naidu KM, Bolliger CT, Diacon AH. Risk factors for recurrence of haemoptysis following bronchial artery embolisation for life-threatening haemoptysis. Int J Tuberc Lung Dis. 2007 Aug;11(8):909-14. PMID 17705959
- [Background] Gross AM, Diacon AH, van den Heuvel MM, Janse van Rensburg J, Harris D, Bolliger CT. Management of life-threatening haemoptysis in an area of high tuberculosis incidence. Int J Tuberc Lung Dis. 2009 Jul;13(7):875-80. PMID 19555538
- [Background] Freitag L, Tekolf E, Stamatis G, Montag M, Greschuchna D. Three years experience with a new balloon catheter for the management of haemoptysis. Eur Respir J. 1994 Nov;7(11):2033-7. PMID 7875278
- [Background] Dutau H, Palot A, Haas A, Decamps I, Durieux O. Endobronchial embolization with a silicone spigot as a temporary treatment for massive hemoptysis: a new bronchoscopic approach of the disease. Respiration. 2006;73(6):830-2. doi: 10.1159/000092954. Epub 2006 Apr 21. PMID 16636529